CLINICAL TRIAL: NCT03844854
Title: The Evaluation of the Usefulness of Shear Wave Sonoelastography in the Diagnosis and Monitoring of the Management of Masseter Muscles Disorders in the Course of Temporomandibular Disorders
Brief Title: Shear Wave Sonoelastography in the Diagnosis and Management of the Masseter Muscles Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wroclaw Medical University (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Anna Olchowy, Principal Investigator, Wroclaw Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PREL.B160.18.007.
Record Dates: First submitted 2018-10-18; First posted 2019-02-19 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Temporomandibular Disorders
Keywords: Sonoelastography; Elastography; Shear-wave; Masseter muscle; Temporomandibular disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: The aim of the first stage is a development of the sonoelastography methodology with precise determination of the positioning of the sonography head and the patient's condyle in temporomandibular joints as well as a determination of the normal range of masticatory muscle structure in the population of healthy subjects. This stage includes people without a history of temporomandibular disorders.
  The second stage is devoted to the assessment of the sonoelastography in the monitoring of the efficacy of treatment. The study group will undergo treatment of masticatory muscles disorders using manual therapy and stabilization occlusal splint. The assessment of severity of pain with Numerical Rating Scale (NRS) and quality of life associated with oral health using standardized international questionnaire will be conducted at baseline and after 12 weeks of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Without intervention.
- Research Group (Experimental): With providing stabilization occlusal splint and manual therapy.
  Interventions: Other: Stabilization occlusal splint and manual therapy

INTERVENTIONS:
Other: Stabilization occlusal splint and manual therapy — Providing stabilization occlusal splint and manual therapy
  Arms: Research Group

SUMMARY:
Contemporary medicine lacks sensitive and objective diagnostic methods for the evaluation of patients with temporomandibular disorders (TMD). Shear wave sonoelastography allows for objective assessment of hardness, tone, and cohesiveness of tissues. Results are expressed in kilopascals (kPa) and can be compared at different time points in the same patient or between patients. The method is non-invasive and safe without any unpleasant experiences for patients.

The project aims to evaluate the usefulness of shear wave sonoelastography in the diagnosis and monitoring of the management of masseter muscles disorders in TMD.

The project will analyze shear wave sonoelastography to determine the pathological tone of masticatory muscles in TMD characterized by pain, abnormal jaw movements and frequent coexistence of headache, otolaryngological disorders, as well as increased tension and pain in the muscles of the neck and shoulder girdle. In the first stage, standardization of sonoelastography of masseter muscles on healthy subjects without TMD will be performed. Normal values of elasticity for various groups of patients as well as factors affecting the result of the study will be determined. Standardization will cover the methodology of the examination. The second stage will assess efficacy of this method in monitoring the treatment progress in patients with TMD diagnosed with the DC-TMD protocol. Standardized sonoelastography examinations and assessment of pain and oral health will be conducted in healthy subjects and in TMD patients at baseline and after 12 weeks of treatment with manual therapy and stabilization occlusal splint. As a result, it will be possible to compare sonoelastography changes in muscle structure in relation to regression of clinical symptoms in response to treatment and to compare sonoelastography results to currently used methods for assessment of TMD.

The need for reliable determining of the sonoelastography values for diagnosis of TMD exist. The hardness of muscles of the human body vary, but norms for masticatory muscles remain undetermined. Available reports are inconclusive. They do not provide a methodology and do not address factors such as age, sex, examination at rest and during jaw-clenching. The present project eliminates those limitations, and as a result, contemporary medicine will get the basis for introducing sonoelastography for the diagnosis and monitoring of masticatory muscles disorders in various groups of patients.

DETAILED DESCRIPTION:
1. Research project objectives/Research hypothesis Masticatory muscles disorders constitute a serious and frequent diagnostic and therapeutic problem in dental practice. Its symptoms appear in 40-90% of the population. The most characteristic symptoms include acute and chronic pain in masticatory muscles and/or temporomandibular joints, sounds in temporomandibular joints (clicking, popping), and abnormal jaw movements. Those main symptoms may be associated with a headache and otolaryngological disorders, as well as increased tension and pain in the muscles of the neck and shoulder girdle. Physical examination shows that masseter muscles disorders are often associated with their hypertrophy and pain during palpation. The pathogenesis of this disorder is unclear and multifactorial. Diagnostic criteria are based on recommendations of INfORM (International Network for Orofacial Pain and Related Disorders Methodology). The main goal of treatment is the elimination of pain in the masticatory muscles.

   The aim of the project is to evaluate the usefulness of shear wave sonoelastography in the diagnosis and monitoring of the progress of treatment of masticatory muscles disorders. To date, few reports attempting to establish normal values have been published, but the available reports have significant limitations.
2. Research project methodology The study is divided into two stages. The aim of the first stage is the development of the sonoelastography methodology with precise determination of the positioning of the sonography head and the patient's condyles in temporomandibular joints as well as the determination of the normal range of masticatory muscle structure in the population of healthy subjects. This stage includes people without the history of TMD and any deviations from normal values according to DC-TMD protocol. Patients treated with drugs affecting masticatory muscles function as well as those with systemic diseases which affect muscle function (e.g., neurological and hormonal disorders, neoplastic disease), above 60 years of age, patients with mental disorders and not agreeing to participate in the study will be excluded.

   Measurement of the masticatory muscle structure will be performed based on the shear wave sonoelastography (SWE) used in the noninvasive assessment of soft tissue hardness. In this method, share waves generated by pressure are detected by longitudinal ultrasonography waves which propagate in the tissues much faster than shear waves. The measurement reflects the quantitative measurement of tissue hardness expressed in kilopascals. Among its advantages are low dependence on the operator, high repeatability and the possibility of quantitative evaluation of tested parameters. The main disadvantage of this method is the fact that every organ has its unique characteristics and hence, normative values must be determined separately for each of them. Examination of masticatory muscles will be conducted by one experienced operator in the same conditions using the same head and the same device. During the examination, the patients will lie on the bed in a supine position. Both masseter muscles will be examined in jaw bite and rest positions.

   The second stage concerning the evaluation of the sonoelastography in the monitoring of the efficacy of treatment. Patients with temporomandibular disorders classified as group II - Masticatory Muscle Disorders (DC-TMD). Exclusion criteria will include previous treatment for masticatory muscles disorders and clinical criteria used in the first stage. Control group will include patients without temporomandibular disorders. The treated group will undergo treatment for masticatory muscles disorders with manual therapy and stabilization occlusal splint. The assessment of severity of pain with Numerical Rating Scale and quality of life associated with oral health using standardized international questionnaire - the Oral Health Impact Profile-14 (OHIP-14) will be conducted at baseline and after 12 weeks of treatment. Masticatory muscle structure as measured with sonoelastography and the results of DC-TMD protocols will be compared in order to evaluate treatment efficacy.
3. Expected impact of the research project on the development of science The investigators expect that the investigator's study will have a large and multidirectional impact on the development of science and the health of society. Gaining reliable method of masticatory muscle structure measurement in the course of masticatory muscles disorders will facilitate the conduct of clinical research by delivering an objective method for comparison of results of treatment conducted in various centers with various methods. The project is also important for public health. Better diagnosis and monitoring of the treatment of this chronic disorder gives a chance for improving oral health care for the entire population. Among the additional values of the project is the interdisciplinarity which is based on the use of cutting-edge non-invasive diagnostic imaging method in oral medicine.

ELIGIBILITY:
Inclusion Criteria:

* First stage with include people without the history of temporomandibular disorders and without any deviations from normal values according to DC-TMD protocol
* Second stage: Patients with TMD without previous history of treatment
* Age between 18 and 60

Exclusion Criteria:

* Patients treated with drugs affecting muscle function
* Not agreeing to participate in the study
* Age under 18
* Age over 60
* Terminal general diseases
* Severe mental disorders
* Neoplasm disease
* Neuromuscular disorders
* Severe hormonal disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-04-20 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Determination of normal elasticity values of the masseter muscle | 12 months
  Elasticity values of the masseter muscle will be measured using shear wave elastography in patients without temporomandibular disorders.
Comparison of elasticity values of the masseter muscle between study groups. | 12 months
  Elasticity values of the masseter muscle will be measured using shear wave elastography in patients with temporomandibular disorders.

SECONDARY OUTCOMES:
Comparison of the mean intensity of pain between study groups. | 12 months
  Pain will be measured with the Visual Analogue Scale (VAS) for pain and reordered before and after the treatment with stabilization occlusal splint and manual therapy. This is a self-reported single-item scale. Patients select a point between 0 score (no pain) and 10 scores (the worst pain ever) on a 10-point scale.
Comparison of oral health status between study groups. | 12 months
  Oral health status will be measured with the Oral Health Impact Profile-14 (OHIP-14) score will be reordered before and after the treatment with stabilization occlusal splint and manual therapy. OHIP-14 consists of 14 items testing 7 domains: functional limitations, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. Response for each question is scored from 0 (the lowest score) to 4 (the highest score). The total scores are calculated by summing response codes. Higher scores indicate poorer oral health status.
Number of participants with treatment-related adverse events | 12 months
  The information about adverse events according to CTCAE v4.0 of the standardised shear wave sonoelastography will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Mieszko Wieckiewicz, DMD MSc PhD, Study Director — Department of Experimental Dentistry, Wroclaw Medical University, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.

REFERENCES:
- [Derived] Olchowy A, Seweryn P, Olchowy C, Wieckiewicz M. Assessment of the masseter stiffness in patients during conservative therapy for masticatory muscle disorders with shear wave elastography. BMC Musculoskelet Disord. 2022 May 11;23(1):439. doi: 10.1186/s12891-022-05392-9. PMID 35546396